CLINICAL TRIAL: NCT03919383
Title: Phase II of Lenvatinib Plus Toripalimab Advanced Hepatocellular Carcinoma: a Single-arm Prospective Trial
Brief Title: Phase II of Lenvatinib Plus Toripalimab for Advanced HCC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Shi Ming, Proffessor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: hcc-S052b
Record Dates: First submitted 2019-04-15; First posted 2019-04-18 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Lenvatinib; Toripalimab
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lenvatinib Plus Toripalimab (Experimental): Participants received lenvatinib capsules 12 milligram (mg) based on the participant's body weight greater than or equal to (>=) 60 kilogram (kg) or 8 mg based on the participant's body weight less than (<) 60 kg at baseline, orally, once daily (QD) in continuous 21-day treatment cycles, and received 240mg toripalimab intravenously every 3 weeks up to documented disease progression, development of unacceptable toxicity, participant request, or withdrawal of consent.
  Interventions: Drug: Lenvatinib; Drug: Toripalimab

INTERVENTIONS:
Drug: Lenvatinib — 12 mg (or 8 mg) once daily (QD) oral dosing
Drug: Toripalimab — 240mg intravenously every 3 weeks

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of lenvatinib combined with toripalimab in patients with advanced hepatocellular carcinoma (HCC)

DETAILED DESCRIPTION:
Lenvatinib was non-inferior to sorafenib in overall survival in untreated advanced hepatocellular carcinoma. No study has evaluated the efficacy and safety of lenvatinib plus toripalimab. Thus, the investigators carried out this single-arm, prospective, phase II study to find out it.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of HCC was based on the diagnostic criteria for HCC used by the European Association for the Study of the Liver (EASL)
* Patients must have at least one tumor lesion that can be accurately measured according to EASL criteria.
* Barcelona clinic liver cancer-stage C
* Eastern Cooperative Oncology Group performance status of 0 to 2
* with no previous systemic treatment
* No Cirrhosis or cirrhotic status of Child-Pugh class A only
* Not amendable to surgical resection ,local ablative therapy and any other cured treatment.
* The following laboratory parameters:

Platelet count ≥ 75,000/μL Hemoglobin ≥ 8.5 g/dL Total bilirubin ≤ 30mmol/L Serum albumin ≥ 30 g/L ASL and AST ≤ 5 x upper limit of normal Serum creatinine ≤ 1.5 x upper limit of normal INR ≤ 1.5 or PT/APTT within normal limits Absolute neutrophil count (ANC) >1,500/mm3 Ability to understand the protocol and to agree to and sign a written informed consent document

Exclusion Criteria:

* Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
* Known history of HIV
* History of organ allograft
* Known or suspected allergy to the investigational agents or any agent given in association with this trial.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Evidence of bleeding diathesis.
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* Known central nervous system tumors including metastatic brain disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
6 months progression free survival rates | 6 months
  Progression was defined as progressive disease by independent radiologic review according to RECIST, version 1.1, criteria or death from any cause.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 6 months
  PFS was defined as the time from the date of randomization to the date of first documentation of disease progression based on Response Evaluation Criteria in Solid Tumors (RECIST), or date of death, whichever occurred first.
Overall Survival (OS) | 6 months
  OS was defined as the duration from the date of randomization until the date of death from any cause. Participants who were lost to follow-up were censored at the last date the participant was known to be alive, and participants who remained alive were censored at the time of data cutoff.
Objective Response Rate (ORR) | 6 months
  ORR was defined as the percentage of participants with a best overall response of complete response (CR) or partial response (PR) based on RECIST. CR was defined as disappearance of any intratumoral arterial enhancement in all target lesions. PR was defined as at least a 30% decrease in the sum of diameters of viable (enhancement of arterial phase) target lesions taking as reference to the baseline sum of the diameters of target lesions
Adverse Events | 6 months
  Number of adverse events. Postoperative adverse events were graded based on CTCAE v4.03

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center Sun Yat-sen University, Guangzhou, Guangdong, China